CLINICAL TRIAL: NCT00071279
Title: The Van Gogh-extension Trial, a Multicenter, International, Randomized, Double-blind, Study Comparing the Efficacy and Safety of Once-weekly Subcutaneous SR34006 With Placebo in the Long-term Prevention of Symptomatic Venous Thromboembolism in Patients With Symptomatic Pulmonary Embolism or Deep-vein Thrombosis Who Completed 6 Months of Treatment With Vitamin K Antagonist or SR34006
Brief Title: SR34006 Compared to Placebo in Patients Who Have Completed 6 Months of Treatment for Symptomatic Pulmonary Embolism or Deep Vein Thrombosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Masking: Double
Other Study IDs: EFC5135; SR34006
Record Dates: First submitted 2003-10-16; First posted 2003-10-20 (Estimated); Last update posted 2011-04-06 (Estimated); Status verified 2011-04

CONDITIONS: Pulmonary Embolism; Deep Vein Thrombosis
MeSH Terms: conditions — Pulmonary Embolism; Venous Thrombosis | interventions — idraparinux; Injections

INTERVENTIONS:
Drug: SR34006 (idraparinux sodium) Injection

SUMMARY:
Patients diagnosed with pulmonary embolism (blood clot in the lung) or deep vein thrombosis (blood clot in a leg vein) are at risk for these blood clots to reoccur. Anticoagulant (blood-thinning) drugs are normally given immediately after the clot is discovered and are continued for a period of 3 or 6 months during which time the risk for recurrence is highest. Research has shown that when oral anticoagulants are used appropriately during this period, patients are less at risk for a recurrent blood clot and this risk reduction outweighs the potential for bleeding to occur.

In this study, patients who had a blood clot in the lung or in a leg vein and completed 6 months of treatment with daily oral vitamin K antagonists (acenocoumarol or warfarin) or once-weekly injections of SR34006 (a new anticoagulant drug) will receive an additional 6 months of once-weekly SR34006 injections or injections of a solution containing no drug (placebo). This trial will evaluate whether patients treated for an additional 6 months with SR34006 have fewer recurrences of blood clots when compared to patients treated with placebo.

Assignment to either SR34006 or placebo will be purely by chance. Neither the patients nor their doctors will know which treatment is being given.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed symptomatic Pulmonary Embolism (PE) or Deep Vein Thrombosis (DVT) who have been treated with acenocoumarol, warfarin or SR34006 for six months
* Written informed consent

Exclusion Criteria:

* Legal age limitations (country specific)
* Indication for anticoagulation other than PE or DVT
* Creatinine clearance (CLcr) <10 mL/min, severe hepatic disease, or bacterial endocarditis
* Participation in a pharmacotherapeutic study other than the Van Gogh-PE or DVT study within the prior 30 days
* Life expectancy <3 months
* Patients in whom anticoagulation treatment for their index PE or DVT should be continued beyond 6 months
* Active bleeding or high risk for bleeding
* Uncontrolled hypertension: systolic blood pressure >180 mm Hg or diastolic blood pressure > 110 mm Hg
* Pregnancy, or childbearing potential without proper contraceptive measures, women who are breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1215 (Actual)
Dates: Start 2003-11; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Symptomatic recurrent PE/DVT during the 6-month study treatment period.

SECONDARY OUTCOMES:
Major bleeding during the 6-month study treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (65):
- United States (32):
  - Bay Pines VA Medical Center, Bay Pines, Florida
  - Pulmonary Associates of Brandon, Brandon, Florida
  - Jacksonville Cardiovascular Clinic, Jacksonville, Florida
  - Melbourne Internal Medicine Associates (MIMA), Melbourne, Florida
  - Melbourne Internal Medical Associates (MIMA), Palm Bay, Florida
  - Clinical Pharmacology Services, Tampa, Florida
  - Medical College of Georgia, Augusta, Georgia
  - Cardinal Bernardin Cancer Center, Maywood, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Dr. Kiritkumar C. Patel's and Dr. Michele DeGregorio's Office, Bloomfield Hills, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - St. Joseph Mercy - Oakland Clinical Research Office, Pontiac, Michigan
  - St. Joseph Mercy - Oakland, Pontiac, Michigan
  - William Beaumont Hospital / Clinical Research Center, Royal Oak, Michigan
  - William Beaumont Hospital Troy, Troy, Michigan
  - Lovelace Sandia Health Systems, Clinical Thrombosis Center, Albuquerque, New Mexico
  - University of New Mexico Hospital, Albuquerque, New Mexico
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Crozer-Chester Medical Center, Upland, Pennsylvania
  - Lung & Chest Medical Associates, Spartanburg, South Carolina
  - Spartanburg Pharmaceutical Research, Spartanburg, South Carolina
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - The Methodist Hospital, Houston, Texas
  - Scott and White Memorial Hospital and Clinic, Temple, Texas
  - The University of Texas Health Center at Tyler, Tyler, Texas
  - Inova Alexandria Hospital, Alexandria, Virginia
  - Pulmonary Associates of Fredericksburg, Inc., Fredericksburg, Virginia
  - McGuire VA Medical Center, Richmond, Virginia
  - Swedish Medical Center, Seattle, Washington
  - Pulmonary Specialists/Spokane Respiratory Consultants, Spokane, Washington
  - Sacred Heart Medical Center, Spokane, Washington
- Australia (3):
  - Box Hill, Clayton, Coffs Harbour, Garran, Kogarah
  - Premantle, Redcliffe, Saint Leonards, South Australia
  - Ringwood East, Woolloongabba
- Graz, Wien, Austria
- Bruxelles, Duffel, Leuven, Lier, Zottegem, Belgium
- Porto Alegre, Salvador, Sao Paulo, Brazil
- Canada (7):
  - University of Alberta, Edmonton, Alberta
  - Kelowna General Hospital, Kelowna, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - The Ottawa Hospital, Civic Campus, Ottawa, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - Centre hospitalier de l'Universite Laval du Centre hospitalier universitaire de Quebec, Sainte-Foy, Quebec
- Czechia (2):
  - Brno, Hradec Karlove, Jihlava, Karlovy Vary, Kladno
  - Ostrava-Poruba, Plzen, Prague, Usti Nad Labem
- Denmark (2):
  - Arhus, Braedstrup, Frederiksberg, Glostrup, Hillerod
  - Kobenhavn, Odense
- Seinäjoki, Finland
- France (3):
  - Besancon, Brest, Chambray Les Tours, Clamart, Grenoble
  - Montpellier, Paris, Rouen, Saint Brieuc, Saint Etienne
  - Toulouse, Valenciennes
- Berlin, Bochum, Dresden, Heidelberg, Ibbenburen, Mannheim, Germany
- Italy (2):
  - Genova, Milano, Padova, Parma, Pavia, Piacenza, Reggio Emilia
  - Treviso, Venezia
- Netherlands (2):
  - Alkmaar, Almere, Amersfoort, Amsterdam, Arnhem, Haarlem
  - Maastricht, Nieuwegein, Sittard, Zwolle
- Auckland, New Zealand
- Oslo, Rud, Norway
- Bialystok, Szczecin, Warszawa, Wroclaw, Poland
- Bloemfontein, Bryanston, Durban, South Africa
- Barcelona, Madrid, Torrelavega, Xativa, Spain
- Goteborg, Jonkoping, Stockholm, Varnamo, Vastervik, Sweden
- London, United Kingdom

REFERENCES:
- [Derived] van Gogh Investigators; Buller HR, Cohen AT, Davidson B, Decousus H, Gallus AS, Gent M, Pillion G, Piovella F, Prins MH, Raskob GE. Extended prophylaxis of venous thromboembolism with idraparinux. N Engl J Med. 2007 Sep 13;357(11):1105-12. doi: 10.1056/NEJMoa067703. PMID 17855671
- See also: Related Info — http://www.sanofi-aventis.com